CLINICAL TRIAL: NCT05253261
Title: Decompression of Odontogenic Cysts Using an Appliance Fabricated With a Fully Digital Workflow
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Marton Kivovics, Head of the Oral Surgery Unit, Semmelweis University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020/109DD
Record Dates: First submitted 2022-02-15; First posted 2022-02-23 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Odontogenic Cysts
Keywords: 3D printing; rapid prototyping; decompression; enucleation; cystostomy
MeSH Terms: conditions — Odontogenic Cysts | interventions — Radionuclide Imaging; Tooth Extraction; Cystostomy; Decompression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Odontogenic cyst treated by decompression with an appliance. (Experimental): Cystostomy procedure is carried out with the same day delivery of a decompression appliance fabricated with a fully digital workflow. Enucleation of the cyst is carried out following decompression.
  Interventions: Diagnostic Test: Preoperative Cone Beam Computed Tomography (CBCT) scan; Procedure: tooth removal and cystostomy; Procedure: Decompression; Diagnostic Test: Postoperative Cone Beam Computed Tomography (CBCT) scan; Procedure: Cyst Enucleation

INTERVENTIONS:
Diagnostic Test: Preoperative Cone Beam Computed Tomography (CBCT) scan — CBCT scans (Green X, Vatech, Hwaseong, Korea) are carried out prior to cystostomies. The scanning conditions are constant at 200 µm isotropic voxel size with 360° rotation, 94 kV tube voltage, 7.2 mA tube current and 9 s exposure time with a 15 × 8 cm field of view field of view (FOV).
Procedure: tooth removal and cystostomy — Surgical interventions are carried out in local anaesthesia. If it is deemed that a tooth or teeth included in the odontogenic cyst is of hopeless prognosis, it is removed at the time of cystostomy procedure. During cystostomy a bony window is created to accessthe cyst. The lining of the cyst is opened to accomodate the tube of the decompression appliance. A sample from the lining of the cyst is sent for histologic evaluation to confirm the diagnosis of odontogenic cyst.
Procedure: Decompression — The decompression appliances is delivered in the same sitting as the cystostomy. Patients are instructed on how to wear and clean their decompression device and are recalled for clinical examinations.
Diagnostic Test: Postoperative Cone Beam Computed Tomography (CBCT) scan — Postoperative CBCT examination is performed six months into the decompression period using the same scanning conditions as those used for the preoperative CBCT scan.
Procedure: Cyst Enucleation — Following the decompression period enucleation of the remaining cyst is carried out in local anaesthesia.

SUMMARY:
The aim of this prospective case series is to present clinical results with cystostomy, decompression and final enucleation of odontogenic cysts using a decompression device fabricated with a full digital workflow and delivered on the day of cystostomy. The secondary purpose of our study is to present the volumetric changes of the odontogenic cysts treated by decompression.

DETAILED DESCRIPTION:
Cystostomy and decompression Patients rinse with 0.2% chlorhexidine solution for 1 min before surgery. Under local anesthesia, an envelope flap from marginal incision is elevated and teeth deemed for extraction are removed in an atraumatic manner. In those cases where the cyst may not be accessed from the sockets of the teeth removed osteotomies are carried out by round burs using a surgical handpiece (SURGmatic S11 L Pro , Kavo Dental, Brea, California, United States) and motor (MASTERsur LUX, Kavo Dental, Brea, California, United States) to create a bony window. A histological sample is collected from the cyst lining to confirm the initial diagnosis of odontogenic cyst. Wound margins are stabilized using single interrupted sutures. The decompression appliance is delivered in the same sitting. Patients are instructed on how to wear and clean their decompression device. Antibiotics (1 g amoxicillin-clavulanate twice a day for 5 days or, in case of side effects or known allergy to penicillin, 300 mg clindamycin 4 times a day for 4 days), non-steroid anti-inflammatory drugs (50 mg diclofenac 3 times a day for 3 days), and chlorhexidine mouthwash (twice a day for 21 days from the first day after surgery) are prescribed. Sutures are removed after 7 days

Postoperative imaging Postoperative CBCT examination is performed six months into the decompression period using the same scanning conditions as those used for the preoperative CBCT scan.

Data acquisition Pre- and postoperative CBCT reconstructions are registered by landmark registration using the 3DSlicer 4.10.2 (The Brigham and Women's Hospital, Inc., Boston, MA, USA) software. The volume of the odontogenic cysts before (Preoperative Volume) and following (Postoperative Volume) decompression are assessed by manual segmentation using the segment editor and segment statistics plug-in. Volume Reduction is calculated by subtracting the Postoperative Volume from the Preoperative Volume. Percentage of Volume Reduction is calculated as follows: Volume Reduction/Preoperative Volume X 100.

Decompression Decompression is maintained until the cyst reduces in volume to an extent, that enucleation may be performed with minimal risk of complications (damage to the anatomical landmarks blood vessels, nerves, roots of neighboring teeth, nasal cavity, maxillary sinuses). During the decompression period patients are recalled for clinical examination and radiographic control (panoramic radiographs) monthly.

Enucleation Following decompression enucleation of the remaining cyst is carried out under local anaesthesia.

Patients are recalled for clinical examination and radiographic control (panoramic radiographs) a year after enucleation to determine whether recurrence of the odontogenic cyst occurs or not.

ELIGIBILITY:
Inclusion Criteria:

* Patients of the Department of Community Dentistry, Semmelweis University, presenting with odontogenic cysts of the jaws that involved anatomical landmarks were included in the study.

Exclusion Criteria:

* History of tumors or irradiation therapy in the head and neck region,
* History of uncontrolled medical or psychiatric disorders,
* Unwillingness to return for follow-up appointments.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Success of the treatment of the odontogenic cyst by the approach described | Decompression may take at least 6 months up to 18 months and lasts until the enucleation may be carried out with minimal risk of complicatios to anatomical landmarks included in the cyst.
  The odontogenic cyst is resolved clinically and radiologically by bony healing
Recurrence | One year after enucleation
  During follow up recurrence of the odontogenic cyst is observed

SECONDARY OUTCOMES:
Volumetric changes | 6 months to 18 months. The timeframe of decompression.
  Volumetric changes of the cyst cavity during decompression.

CONTACTS AND LOCATIONS:
Overall Officials: Márton Kivovics, DMD MSc PhD, Principal Investigator — Semmelweis University Department of Community Dentistry
Locations (1):
- Semmelweis University Department of Community Dentistry, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kivovics M, Penzes D, Moldvai J, Mijiritsky E, Nemeth O. A custom-made removable appliance for the decompression of odontogenic cysts fabricated using a digital workflow. J Dent. 2022 Nov;126:104295. doi: 10.1016/j.jdent.2022.104295. Epub 2022 Sep 15. PMID 36116543